CLINICAL TRIAL: NCT01271556
Title: Salmeterol Improves Fluid Clearance From Alveolar-Capillary Membrane in COPD Patients
Brief Title: Effect of Salmeterol on Fluid Clearance From Alveolar-Capillary Membrane in COPD Patients
Acronym: SALM1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Dr. Fabiano Di Marco, Respiratory Unit, San Paolo Hospital, University of Milan, Milan, Italy
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SALM101012008
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2008-12

CONDITIONS: Salmeterol Effect Against an Acute Alveolar Fluid Clearance Challenge Secondary to Lung Fluid Overload in COPD Patients; Chronic Obstructive Pulmonary Disease; Bronchodilator Agents; Salmeterol
Keywords: COPD; LABA; salmeterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1, salmeterol, saline infusion (Experimental): In 10 COPD patients and 10 healthy subjects, tiotropium and long-acting and short-acting beta-2 agonists were withdrawn at least 72 hours if assumed, 24 hours, and 12 hours, respectively, prior to each test day. Salmeterol 50 mcg on days A was administered between 8 AM and 10 AM. Patients and healthy subjects underwent a rapid 50-minute 750-ml 0.9% saline infusion 240 minutes after inhalatory treatment (salmeterol 50 mcg MDI), and mixed venous blood was withdrawn for measurements of hematocrit (Htc), Hb, and albumin concentration 10 minutes before and 10 minutes after the infusion. 240 and 290 minutes after inhalatory treatment, pulmonary function tests were performed.
  Interventions: Drug: Salmeterol; Procedure: saline infusion (0.9 per cent sodium chloride)
- 2, placebo, saline infusion (Placebo Comparator): In 10 COPD patients and 10 healthy subjects, tiotropium and long-acting and short-acting beta-2 agonists were withdrawn at least 72 hours if assumed, 24 hours, and 12 hours, respectively, prior to test day. Placebo was administered between 8 AM and 10 AM. Patients and healthy subjects underwent a rapid 50-minute 750-ml 0.9% saline infusion 240 minutes after inhalatory treatment (placeboI), and mixed venous blood was withdrawn for measurements of hematocrit (Htc), Hb, and albumin concentration 10 minutes before and 10 minutes after the infusion. 240 and 290 minutes after inhalatory treatment, pulmonary function tests were performed.
  Interventions: Procedure: saline infusion (0.9 per cent sodium chloride); Other: Placebo
- 3, salmeterol, no saline infusion (Active Comparator): In 10 COPD patients and 10 healthy subjects, tiotropium and long-acting and short-acting beta-2 agonists were withdrawn at least 72 hours if assumed, 24 hours, and 12 hours, respectively, prior to test day. Salmeterol 50 mcg on days A was administered between 8 AM and 10 AM. 240 and 290 minutes after inhalatory treatment, pulmonary function tests were performed.
  Interventions: Drug: Salmeterol
- 4, placebo, no saline infusion (Placebo Comparator): In 10 COPD patients and 10 healthy subjects, tiotropium and long-acting and short-acting beta-2 agonists were withdrawn at least 72 hours if assumed, 24 hours, and 12 hours, respectively, prior to test day. Placebo was administered between 8 AM and 10 AM. 240 and 290 minutes after inhalatory treatment (placebo), pulmonary function tests were performed.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Salmeterol — 50 mcg MDI (inhalatory), once on days A and C at t=0,
  Other Names: long acting bronchodilator agents
  Arms: 1, salmeterol, saline infusion; 3, salmeterol, no saline infusion
Procedure: saline infusion (0.9 per cent sodium chloride) — rapid 50-minute 750-ml 0.9% saline infusion 240 minutes after inhalatory treatment on day A and B
  Other Names: physiologic saline solution
  Arms: 1, salmeterol, saline infusion; 2, placebo, saline infusion
Other: Placebo — placebo, inhalatory (MDI) once
  Arms: 2, placebo, saline infusion; 4, placebo, no saline infusion

SUMMARY:
The cardiovascular component associated with COPD plays a major role in prognosis of the disease, being responsible of 25% of the deaths. Experimental and initial clinical data suggest that beta-adrenergic agonists accelerate clearance of excess fluid from the alveolar airspace, with potential positive effect on cardiogenic pulmonary edema.

The aim of this study was to investigate the effects of a long-acting beta-2 agonist, salmeterol, on alveolar fluid clearance in COPD patients by evaluating the diffusive and mechanical lung properties. Our experimental model to test alveolar fluid clearance was rapid saline intravenous infusion.

Ten COPD and 10 healthy subjects treated with salmeterol or placebo 4 hours before the begin of the study were evaluated, in four non consecutive days, just before and after a saline infusion or a similar period without infusion.

Both in COPD and healthy subjects rapid saline infusion, with placebo or salmeterol premedication, lead to a significant decrease of DLCO and FEV1. Nonetheless, salmeterol pretreatment lead to a significant reduction of the impairment of gas exchange due to saline infusion (-64% of DLCO reduction in comparison with placebo), whilst it did not affect the changes in FEV1. In the control setting, with no infusion, we did not find any significant change of both DLCO and mechanical properties of the lung.

In conclusions, in COPD patients salmeterol appears to provide a protective effect against an acute alveolar fluid clereance challenge secondary to lung fluid overload providing an intriguing mechanistic explanation for the benefits observed in larger trials.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis (consistent with the diagnostic standards of the European Respiratory Society, ERS, for the management of COPD)
* stable condition for ≥4 weeks and had a prebronchodilator forced expiratory volume in one second (FEV1) of <60% of the predicted value

Exclusion Criteria:

* known allergies to the study medication
* long-term oxygen therapy
* history of asthma, allergic rhinitis, atopy, or a total blood eosinophil count greater than 400/mm3
* chronic heart failure, untreated arterial hypertension, myocardial infarction within the last 6 months, diabetes mellitus
* increased serum potassium levels.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
change caused by the effect of salmeterol on lung diffusion capacity for carbon monoxide (DLCO) and its components after a challenge with rapid intravenous saline infusion | 240 and 290 minutes after inhalatory treatment pulmonary function tests were performed
  DLCO was measured twice (Sensor Medics 2200 Pulmonary Functional Test System, USA) for each oxygen mixture, with washout intervals of at least 4 minutes (the average was taken as the final result), according to the European Respiratory Society guidelines. The single-breath alveolar volume (VA) was derived by methane dilution. Alveolar-capillary membrane diffusing capacity (DM) and capillary blood volume available for gas exchange (Vc) were determined with the same equipment, according to the classic Roughton and Forster method

SECONDARY OUTCOMES:
changes in mechanical lung properties | 240 and 290 minutes after inhalatory treatment
  Mouth flow was measured by a mass flowmeter, and volume was obtained by numerical integration of the flow signal. Spirometry and flow-volume curves were obtained by manoeuvres consisting of six to eight regular tidal breaths, a forced expiration initiated from end-tidal inspiration to residual volume (partial expiratory flow-volume curve, PEFV), followed by a fast inspiration to total lung capacity and a forced expiration to residual volume (maximal expiratory flow-volume curve, MEFV).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Centanni, MD, Study Director — Respiratory Medicine Section, Dipartimento Toraco-Polmonare e Cardiocircolatorio, Università degli Studi di Milano, San Paolo Hospital
Locations (1):
- Respiratory Medicine Section, Dipartimento Toraco-Polmonare e Cardiocircolatorio, Università degli Studi di Milano, San Paolo Hospital, Milan, Milan, Italy